CLINICAL TRIAL: NCT07090954
Title: An Open-Label, Multicenter, Phase Ib/II Clinical Trial of GR1803 Injection in Combination With an Anti-CD38 Monoclonal Antibody Evaluating Safety, Pharmacokinetics, Immunogenicity, and Preliminary Efficacy in Subjects With Relapsed/Refractory Multiple Myeloma Previously Treated With at Least One Line of Therapy Including Lenalidomide and a Proteasome Inhibitor
Brief Title: A Study of GR1803 Injection in Combination With Anti-CD38 Monoclonal Antibody for the Treatment of Participants With Multiple Myeloma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genrix (Shanghai) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GR1803-003
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GR1803 plus anti-CD38 monoclonal antibody (Experimental): Participants will be assigned to a combination of anti-CD38 monocloncal antibody plus GR1803 injection.
  Interventions: Drug: GR1803 injection; Drug: Anti-CD38 Monoclonal Antibody

INTERVENTIONS:
Drug: GR1803 injection — Participants will receive GR1803 injection.
Drug: Anti-CD38 Monoclonal Antibody — Participants will receive anti-CD38 monoclonal antibody.

SUMMARY:
The purpose of this study is to identify recommended Phase 3 doses (RP3D) for treatment combination (GR1803 injection plus anti-CD38 monoclonal antibody) and to characterize the efficacy of RP3D for the treatment combination.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group performance status grade of 0, 1 or 2;
* Diagnosis of multiple myeloma；have received at least one prior line of therapy including Lenalidomide and a proteasome inhibitor.
* Able to understand and comply with the requirements of the clinical protocol, voluntarily participate in the clinical trial, and sign informed consent.

Exclusion Criteria:

* Plasma cell leukemia , Waldenström's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes), or amyloidosis.
* Active central nervous system involvement or exhibits clinical signs of meningeal involvement of multiple myeloma.
* Prior treatment with any BCMA-targeted therapiy.
* Active infecion.
* Known allergies, hypersensitivity, or intolerance to the study drug or its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation: Number of Participants With Dose Limiting Toxicity (DLT) | Up to 2 Years
  The dose limiting toxicities are defined as any of the following events: drug related hematological or non-hematological toxicity of grade 3 or higher.
Dose escalation: Number of Participants With Adverse Events and Serious Adverse Events | Up to 2 Years
  Adverse event is any untoward medical occurrence in a clinical trial participants administered a pharmaceutical product, regardless of causal relationship to the study treatment. This includes any unfavorable or unintended sign, symptom, or disease temporally associated with the use of the product.
  Serious adverse event is an adverse event that results in any of the following outcomes: death, life-threatening, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, other medically important events.
Dose expansion: Overall Response Rate | Up to 2 Years
  The percentage of participants who have a partial response or better according to the International Myeloma Working Group criteria

SECONDARY OUTCOMES:
Duration of Response | Up to 2 Years
  Time from initial partial response or better to progressive disease or death due to any cause
Progression-Free Survival | Up to 2 Years
  Time from first administration of GR1803 injection to tumor progerssion or death from any cause
Serum Concentration of GR1803 Injection | Up to 2 Years
  Serum concentration of GR1803 injection will be assessed
Number of Participants With Anti-Drug Antibodies to GR1803 Injection | Up to 2 Years
  Number of participants with anti-drug antibodies to GR1803 injection will be assessed

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai Fourth People's Hospital Affiliated with Tongji University, Shanghai
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an